CLINICAL TRIAL: NCT00452777
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group Study Evaluating the Efficacy and Tolerability of Oral BVT.115959, a Novel A2A Agonist, Versus Placebo in the Treatment of Diabetic Neuropathic Pain
Brief Title: Efficacy and Tolerability of Novel A2A Agonist in Treatment of Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVT.115959-005
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Neuropathic Pain
Keywords: Diabetic neuropathy, painful; Adenosine A2A receptor
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BVT.115959 (Experimental): Capsules containing 7 mg BVT.115959 administered orally three times daily
  Interventions: Drug: BVT.115959
- Placebo (Placebo Comparator): Placebo capsules administered orally three times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BVT.115959
  Arms: BVT.115959
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of BVT.115959 in diabetic patients with neuropathic pain who are either not on analgesia or are on stable analgesia in the month prior to entering the study.

DETAILED DESCRIPTION:
The planned study is an exploratory study which aims to provide proof of the efficacy of BVT.115959 in the reduction of the symptoms of pain. Thus, the primary objective is to evaluate the anticipated analgesic properties of BVT.115959 in patients with diabetic neuropathic pain and to confirm its activity against placebo.

The study will evaluate the efficacy and tolerability of oral BVT.115959 7 mg administered three times a day (t.i.d.) versus a matching placebo in diabetic patients with neuropathic pain who are either not on analgesia or are on stable analgesia in the month prior to entering the study and who are being maintained on stable analgesia throughout the study. Eligible subjects will be randomized in a ratio of 2:1 (BVT.115959: placebo).

The study consists of a 1-week screening/baseline period, a 4-week treatment period and a 1 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 1 or 2 diabetes mellitus and documented painful, symmetrical, sensorimotor polyneuropathy for at least 6 months
* Either no analgesic medication or on stable analgesic medication for at least 4 weeks

Exclusion Criteria:

* Female patients who are fertile and of child-bearing potential
* Clinically significant or unstable hepatic, respiratory, renal, hematologic, cardiovascular or peripheral vascular disease
* Painful conditions that may confound the evaluation of neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in mean 24-hour pain intensity score from baseline using an 11-point Likert NRS assessed over the preceding 24 hours immediately upon awakening in the morning

SECONDARY OUTCOMES:
Present pain intensity using an 11-point Likert NRS assessed at bedtime
Short-Form McGill Pain Questionnaire parameters
Weekly mean sleep interference score
Clinical Global Impression of Change and Patient's Global Impression of Change
Quality of life
Mood stability
Time to study withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Keith Bragman, MD FRCP FRCPath FFPM, Study Director — Swedish Orphan Biovitrum
Locations (20):
- Czechia (4):
  - Biovitrum investigational site, České Budějovice
  - Biovitrum investigational site, Litoměřice
  - Biovitrum investigational site, Pilsen
  - Biovitrum investigational site, Prague
- Germany (8):
  - Biovitrum Investigational Site, Bad Kreuznach
  - Biovitrum Investigational Site, Berlin
  - Biovitrum Investigational Site, Dortmund
  - Biovitrum Investigational Site, Gelsenkirchen
  - Biovitrum Investigational Site, Hamburg
  - Biovitrum Investigational Site, Mainz
  - Biovitrum Investigational Site, Mannheim
  - Biovitrum Investigational Site, Neumünster
- South Africa (8):
  - Biovitrum Investigational Site, Bloemfontein
  - Biovitrum Investigational Site, Durban
  - Biovitrum Investigational Site, Kenilworth
  - Biovitrum Investigational Site, Kraaifontein
  - Biovitrum Investigational Site, Polokwane
  - Biovitrum Investigational Site, Pretoria
  - Biovitrum Investigational Site, Somerset West
  - Biovitrum Investigational Site, Wynberg